CLINICAL TRIAL: NCT07137923
Title: Single Maintenance And Reliever Therapy Strategies for IMPLementation and Effectiveness (SMART & SIMPLE) Trial
Brief Title: SMART Implementation-Effectiveness Trial 1
Acronym: SMART & SIMPLE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 23-021702 A; R01HL173600 (NIH)
Record Dates: First submitted 2025-08-15; First posted 2025-08-22 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Asthma in Children
MeSH Terms: interventions — Educational Status

STUDY DESIGN:
Intervention Model Description: This study will use a cluster randomized control trial (RCT) study design to test the impact of the clinical decision support and education (CDS+) to increase adoption of SMART therapy.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Clinics in Arm 1 will receive the intervention in Interval 1. Interval 1 intervention: clinical decision support and education (CDS+).
  Interventions: Behavioral: Clinical decision support + education (CDS+)
- Control (Active Comparator): Clinics in Arm 2 will not be exposed to the interventions.
  Interventions: Other: Control

INTERVENTIONS:
Behavioral: Clinical decision support + education (CDS+) — Intervention clinic providers will experience nudges in the electronic medical record to encourage prescribing SMART where clinically-appropriate and intervention clinic providers, families/patients, and nurses will receive education (collectively CDS+).
  Other Names: CDS+
  Arms: Intervention
Other: Control — Clinics in Arm 2 will not be exposed to the interventions.
  Arms: Control

SUMMARY:
While single maintenance and reliever therapy (SMART) has been the preferred management strategy for Step 3 and 4 (moderate/severe) asthma management since the 2020 NIH asthma guideline updates, adoption of SMART has not been rigorously assessed. This study will test electronic medical record clinical decision support and education implementation strategies (CDS+) to increase adoption of SMART in pediatric primary care. This is the first of two related records.

DETAILED DESCRIPTION:
Asthma is a leading cause of childhood morbidity nationwide. Limited provider adoption of and patient adherence to the prevailing evidence-based recommendations for chronic management represent tractable areas for care improvement and implementation focus. In their 2020 Focused Updates, the NHLBI codified a new paradigm of asthma management - single maintenance and reliever therapy (SMART) - as the preferred management strategy for Steps 3 and 4 (moderate/severe) asthma management. In addition to its efficacy and safety, SMART has demonstrated real-world effectiveness in international settings, likely due in part to better adherence to daily therapy and less inhaler confusion. However, SMART has not been widely implemented in practice in the U.S. This hybrid type II implementation-effectiveness study will sequentially compare the effects of usual care to (1) electronic health record-based clinical decision support plus education (CDS+) (Study 1 - current study) and then (2) CDS+ with population health management (PHM) strategies (community health worker and nurse care manager) on SMART adoption (Study 2). Randomization for this study is at the clinic-level. Results will be reported at visit-, patient-, and clinic-levels.

ELIGIBILITY:
Clinic Inclusion Criteria:

* The clinic is a pediatric primary care clinic that is part of the Children's Hospital of Philadelphia (CHOP) Pediatric Research Consortium (PeRC).
* The clinic agrees to participate in SMART & SIMPLE study.

Clinic Exclusion Criteria:

- The clinic is not willing to participate in SMART & SIMPLE study interventions.

Patient Inclusion Criteria:

* Ages 5-18 years;
* Has clinic visit at participating practice during study interval (sick, well, or follow-up)
* Prescribed at least one prescription for an inhaled corticosteroid (ICS) or ICS-long-acting beta agonist (ICS-LABA) for maintenance asthma therapy in the past year;
* Evidence of uncontrolled asthma as determined by: (1) uncontrolled Asthma Control Tool score in the past 6 months OR (2) two or more systemic corticosteroids prescribed for an asthma exacerbation in the past 12 months (one occurring in the past 6 months)

Patient Exclusion Criteria:

- Transferred clinics or left the CHOP Pediatric Care Network.

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 18 (Estimated)
Dates: Start 2025-09-03 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2028-02-29 (Estimated)

PRIMARY OUTCOMES:
Change in the Rate of Visit-Level SMART Adoption | Assessment of rates from two study intervals: Interval 0 (baseline; 11 months), Interval 1 (CDS+; 11 months). There will be a one month ramp up period at the start of each study interval (ramp up period data will not be included in analyses).
  The difference in the rate of SMART prescribing (initiation) among eligible primary care visits (i.e., when a child is eligible to start SMART) where SMART is first prescribed (initiated) comparing the first intervention period (Interval 1) and the baseline period (Interval 0). Adoption is visit-level. The denominator represents eligible primary care visits, and the numerator represents visits where SMART is first prescribed (initiated).

SECONDARY OUTCOMES:
Change in the Proportion of Patient-Level SMART Sustainment | Assessment of proportions from two study intervals: Interval 0 (baseline; 11 months), Interval 1 (CDS+; 11 months). There will be a one month ramp up period at the start of each study interval (ramp up period data will not be included in analyses).
  The difference in the proportion of patients who are prescribed (initiated) SMART who continue on SMART for at least 6 months comparing the first intervention period (Interval 1) and baseline period (Interval 0). Sustainment is patient-level. The denominator represents patients who are prescribed (initiated) SMART, and the numerator represents patients who continue on SMART for at least 6 months.

OTHER OUTCOMES:
Change in the Proportion of Clinic-Level SMART Penetration | Assessment of proportions from two study intervals: Interval 0 (baseline; 11 months), Interval 1 (CDS+; 11 months). There will be a one month ramp up period at the start of each study interval (ramp up period data will not be included in analyses).
  The difference in the clinic-level proportion of SMART-eligible patients who are prescribed (initiated) and not subsequently discontinued from SMART by the end of the interval comparing the first intervention period (Interval 1) and the baseline period (Interval 0). Penetration is clinic-level. The denominator represents patients who are SMART-eligible in each interval, and the numerator represents patients who are prescribed (initiated) during the interval and still on SMART at the end of the interval.

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States